CLINICAL TRIAL: NCT06043089
Title: Impact of Beetroot Supplementation on Sports Performance, Prooxidant-antioxidant Balance and Sleep in Athletes
Brief Title: Impact of Beetroot Supplementation in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AWF_MSIT
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Athletes received 7 days of placebo (2 × 70 mL of water with beetroot powder with negligible nitrate content).
  Interventions: Dietary Supplement: Beetroot juice supplementation or placebo
- Beetroot group (Experimental): Athletes received 7 days of beetroot juice (2 × 70 mL of beetroot juice ∼12.9 mmol NO3-; Beet It, James White Drinks, Ipswich, UK).
  Interventions: Dietary Supplement: Beetroot juice supplementation or placebo

INTERVENTIONS:
Dietary Supplement: Beetroot juice supplementation or placebo — Athletes received 7 days of beetroot juice supplementation with nitrate supplementation (2 × 70 mL of beetroot juice ∼12.9 mmol NO3-; Beet It, James White Drinks, Ipswich, UK) or placebo (2 × 70 mL of water with beetroot powder with negligible nitrate content).

SUMMARY:
Several previous studies observed a positive effect of beetroot supplementation on sports performance in athletes, mainly in endurance performance. However, less attention has been paid to its effects on short-duration performance, especially in youth athletes. Moreover, only a few previous investigations performed biochemical analyses, including pro-oxidant balance assessments. It is especially important because chronic nitrate intake might directly cause the production of reactive nitrogen species and reactive oxygen species in other subcellular compartments, leading to more oxidative stress. Additionally, no previous study verified the impact of beetroot intake on sleep.

ELIGIBILITY:
Inclusion Criteria:

* male
* good general health assessed by physician
* highly trained
* written consent to participate

Exclusion Criteria:

* medication or dietary supplements used within the previous month, which could potentially impact the study outcomes
* history of sleep nor neurological disorders
* chronic use (6 months) of any antibacterial mouthwash products.

Ages: 14 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Performance test | 7 days after treatment
  yo-yo intermittent recovery test level 1
Changes in nitrates | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood plasma will be obtained to measure nitrate concentration
Changes in nitrites | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood plasma will be obtained to measure nitrite concentration
Changes in prooxidant status | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood plasma will be obtained to measure total oxidative status
Changes in antioxidant status | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood plasma will be obtained to measure total antioxidant capacity
Changes in oxidative stress index | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  The oxidative stress index will be calculated as the ratio of plasma prooxidant to antioxidant status
Changes in nitrooxidative stress markers | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood plasma will be obtained to measure 3-nitrotyrosine concentration
Changes in protein oxidation | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood plasma will be obtained to measure advanced protein oxidation products concentration
Changes in nucleic acid oxidation | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood plasma will be obtained to measure ox-8-hydroxy-2'-deoxyguanosine (8-OHdG) concentration
Changes in lipids oxidation | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood plasma will be obtained to measure thiobarbituric acid reactive substances concentration
Changes in exercise-induced metabolic acidosis | 1) Before the performance test 2) 3 minutes after the performance test 3) 10 minutes after the performance test 4) 20 minutes after the performance test
  Arterialized blood will be obtained to measure lactate concentration
Objective Sleep - Time in bed | nights 1 - 7 during treatment
  Total time spent in bed during the night assessed by sleep radar
Objective Sleep - Sleep-onset latency | nights 1 - 7 during treatment
  The time it takes from when the athlete intends to go to sleep and actually starts to sleep assessed by sleep radar
Objective Sleep - Total sleep time | nights 1 - 7 during treatment
  Total sleep time obtained from sleep onset to time at wake-up assessed by sleep radar
Objective Sleep - Light sleep | nights 1 - 7 during treatment
  Total amount of time in light sleep assessed by sleep radar
Objective Sleep - Deep sleep | nights 1 - 7 during treatment
  Total amount of time in deep sleep assessed by sleep radar
Objective Sleep - REM sleep | nights 1 - 7 during treatment
  Total amount of time in REM sleep assessed by sleep radar
Objective Sleep - Sleep efficiency | nights 1 - 7 during treatment
  The percentage of total sleep time to lights off and leaving bed assessed by sleep radar

SECONDARY OUTCOMES:
Countermovement jump height | 7 days after treatment
Ball speed velocity | 7 days after treatment
Sprint test (0-20m) | 7 days after treatment
Agility T-test | 7 days after treatment
Maximal isometric handgrip strength | 7 days after treatment
Flanker task | 7 days after treatment
Changes in muscle damage markers | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood serum will be obtained to measure myoglobin concentration
Changes in muscle enzymes activity | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood serum will be obtained to measure creatine kinase activity
Changes in inflammation markers | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood serum will be obtained to measure C-reactive protein concentration
Changes in blood count | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Whole blood will be obtained to measure leukocyte count
Changes in anabolic hormones | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood serum will be obtained to measure testosterone concentration
Changes in catabolic hormones | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood serum will be obtained to measure cortisol concentration
Changes in kidney function markers | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood serum will be obtained to measure creatinine concentration
Changes in the purine metabolism marker | 1) baseline - 2) 7th day of treatment - before the supplementation, 3) 7th day of treatment - before the performance test, 4) 7th day of treatment - immediately after the performance test
  Blood serum will be obtained to measure uric acid concentration
Changes in hemoglobin concentration | 1) Before the performance test 2) 3 minutes after the performance test 3) 10 minutes after the performance test 4) 20 minutes after the performance test
  Arterialized blood will be obtained to measure hemoglobin concentration
Changes in hematocrit | 1) Before the performance test 2) 3 minutes after the performance test 3) 10 minutes after the performance test 4) 20 minutes after the performance test
  Arterialized blood will be obtained to measure hematocrit
Changes in plasma volume | 1) Before the performance test 2) 3 minutes after the performance test 3) 10 minutes after the performance test 4) 20 minutes after the performance test
  The change in plasma volume will be calculated using the hemoglobin and hematocrit results

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Filip-Stachnik, Phd, Principal Investigator — University of Physcial Education in Cracow
Locations (1):
- University School of Physical Education in Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No